CLINICAL TRIAL: NCT03355872
Title: A Randomised, Double-blind, Phase I/II Study to Evaluate the PK, PD, Safety, and Efficacy Between HLX01 and Rituximab in Patients With Moderate to Severe Rheumatoid Arthritis and Inadequate Response to Treatment With DMARDs
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLX01-RA01
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX01 (Experimental)
  Interventions: Drug: HLX01
- Rituximab (Active Comparator)
  Interventions: Drug: HLX01

INTERVENTIONS:
Drug: HLX01 — Biosimilar of Rituximab

SUMMARY:
To compare the PK profiles of HLX01 and Rituximab in Chinese patients with moderate to severe rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, between 18 and 65 years of age, who have a diagnosis of moderately to severely active RA for at least 6 months as defined by at least 6 swollen joints (66 joint count) and at least 6 tender joints (68 joint count) at Screening and Baseline (Day 1), and DAS28-CRP>3.2 at Screening. If a joint has both swollen and tender symptoms, then the joint will be included in both the swollen joints and tender joint categories.
2. Current treatment for RA:

   1. Must be currently receiving and tolerating oral or parenteral MTX therapy at a dose of 10 25 mg per week for at least 12 weeks prior to Day 1. The dose should be stable for at least 4 weeks prior to Day 1. Patients must have had an inadequate response to small molecule or biologic DMARD therapy.
   2. Patients must be willing to receive oral folic acid (at least 5 mg/week or as per local practice) or equivalent during the entire study (mandatory co-medication for MTX treatment).
   3. Inadequate response to biologic DMARDs: anakinra and etanercept must be withdrawn at least 4 weeks prior to Day 1; tocilizumab must be withdrawn at least 12 weeks prior to Day 1; other agents must be withdrawn at least 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
   4. Inadequate response to small molecule DMARDs (other than MTX): Leflunomide must be withdrawn at least 8 weeks prior to Day 1 or a minimum of 2 weeks prior to Day 1 if after 11 days of standard cholestyramine washout. Lower than 400 mg/day of oral hydroxychloroquine or lower than 250 mg/day of oral chloroquine is allowed, but the dose should be stable for at least 12 weeks prior to Day 1 until Week 24 (if hydroxychloroquine or chloroquine have been discontinued, they must have been withdrawn at least 4 weeks prior to Day 1). Other DMARDs must be withdrawn at least 4 weeks prior to Day 1.
   5. Tripterygium wilfordii: ongoing therapy is allowed, but the dose should be stable for at least 12 weeks prior to Day 1 until Week 24; if discontinued, T.wilfordii treatment must have been withdrawn at least 2 weeks prior to Day 1.
   6. If receiving current treatment with oral corticosteroids, the dose must not exceed 10 mg/day prednisolone or equivalent. During the 4 weeks prior to Baseline (Day 1) the dose must remain stable until Week 24; if discontinued, oral corticosteroids must have been withdrawn at least 2 weeks prior to Day 1.
   7. Intra-articular and parenteral corticosteroids are not permitted within 6 weeks prior to Baseline Day 1 and throughout the trial (until Week 24), with the exception of IV administration of 100 mg methylprednisolone 30 minutes prior to each infusion as this is part of the trial procedures.
   8. Any concomitant non-steroidal anti-inflammatory drugs (NSAIDs) must be stable for at least 2 weeks prior to Day 1; if discontinued, NSAIDs must have been withdrawn at least 2 weeks prior to Day 1.
3. Males or females of child-bearing potential must agree to use an acceptable method of contraception for 12 months following completion or discontinuation from the trial (e.g., hormonal contraceptive, patch, intrauterine device, physical barrier).

Exclusion Criteria:

1. ACR functional Class IV or wheelchair/bed bound.
2. Primary or secondary immunodeficiency (history of, or currently active), including known history of human immunodeficiency virus infection and Positive HIV.
3. Active tuberculosis (e.g., chest X-ray images of active tuberculosis); for those who have used TNF-α antagonist or in the opinion of the investigator, QUANTIFERON®-TB GOLD will be tested and the positive patients will be excluded.
4. Congestive heart failure (Class III or IV of New York Heart Association)
5. Interstitial lung disease (except mild).
6. Known allergies to mouse protein or other antibodies.
7. History of cancer including solid tumors, hematologic malignancies, and carcinoma in situ (except participants with previous resected and cured basal or squamous cell carcinoma, cervical atypical dysplasia, or in situ Grade I cervical cancer at least 1 year prior to the Screening Visit).
8. Receipt of a live/attenuated vaccine within 12 weeks prior to the Screening Visit until Week 24.
9. Any disease or treatment (including biotherapy) that may bring unacceptable risk to the subject, in the opinion of the investigator
10. Pregnant or lactating female subjects, or subjects who are planning to conceive or breastfeed during the study period or within 12 months after the last administration.
11. History of, or current, inflammatory joint disease other than RA (e.g., gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease) or other systemic autoimmune disorder (e.g., systemic lupus erythematosus, inflammatory bowel disease, pulmonary fibrosis, or Felty's syndrome, scleroderma, inflammatory myopathy, mixed connective tissue disease, or any overlap syndrome).
12. Evidence of significant uncontrolled concomitant disease such as, but not limited to, nervous system, renal, hepatic, endocrine, or gastrointestinal disorders which, in the investigator's opinion, would preclude patient participation.
13. Positive anti-HCV antibodies at screening.
14. Positive anti-TP antibodies at screening.
15. Positive HBsAg or HBcAb, or HBV DNA ≥1×103 copies/mL at screening.
16. Any active infection (except nail bed fungal infection), or any serious infections needed hospitalized or intravenous anti-infective treatment within 4 weeks before the screening visit; or oral anti-infective therapy within 2 weeks before the screening visit.
17. History of deep gap/tissue infection (e.g. fasciitis, abscess, osteomyelitis) within 52 weeks prior to the screening visit.
18. Experienced serious or opportunistic infection in the recent 2 years in the opinion of the investigator.
19. History of chronic infection (such as chronic pyelonephritis, bronchiectasis or osteomyelitis)
20. Any congenital or acquired neurological disease, vascular disease or systemic disease, especially joint pain and swelling (e.g., Parkinson's disease, cerebral palsy, diabetic neuropathy) that may affect the effects assessment of this study.
21. History of alcohol abuse, drug abuse within 52 weeks prior to the screening visit (judged by the investigator).
22. Received anti-integrin αV antibody or cell depletion therapy within 3 months or 5 half-lives (whichever is longer) prior to the screening visit.
23. Intolerant to glucocorticoid injection or has contraindication to glucocorticoid.
24. AST or ALT >2 times ULN. Or haemoglobin < 8.0 g/dL. Or absolute neutrophil count < 1.5x109/L. Or platelet count < 75x109/L.
25. Participated in any clinical study (within 12 weeks or within 5 half-lives of the study drug, whichever is longer).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
AUC(0-inf) | 24weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ann Rheum Dis 2019, 78, 1140-1140 — http://dx.doi.org/10.1136/annrheumdis-2019-eular.3669
- See also: A new population model validated pharmacokinetic similarity of HLX01 and rituximab in B-cell lymphoma. Annals of Oncology 2019, 30. — https://doi.org/10.1093/annonc/mdz251.015
- See also: 266OA population pharmacokinetic model: Assessment of pharmacokinetic similarity of HLX01 and rituximab in diffuse large B-cell lymphoma. Annals of Oncology 2019, 30 (suppl_9), mdz427. — https://doi.org/10.1093/annonc/mdz427